CLINICAL TRIAL: NCT04417530
Title: A Phase 2 Open-label, Ascending Single and Repeat Dose Escalation Trial of Belzupacap Sarotalocan (AU-011) Via Suprachoroidal Administration in Subjects With Primary Indeterminate Lesions and Small Choroidal Melanoma
Brief Title: Phase 2 Trial to Evaluate Belzupacap Sarotalocan (AU-011) Via Suprachoroidal Administration in Subjects With Primary Indeterminate Lesions and Small Choroidal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AU-011-202
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Uveal Melanoma; Ocular Melanoma; Choroidal Melanoma
Keywords: Uveal Melanoma; Eye Cancer; Ocular Melanoma; Choroidal Melanoma
MeSH Terms: conditions — Uveal Melanoma; Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Cohort 1 AU-011& Laser (Experimental): Low dose of AU-011 + 1 laser application
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser
- Cohort 2 AU-011 & Laser (Experimental): Medium dose of AU-011 + 1 laser application
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser
- Cohort 3 AU-011 (belzupacap sarotalocan) & Laser (Experimental): Medium dose of AU-011 + 2 laser applications
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser
- Cohort 4 AU-011 & Laser (Experimental): Highest tolerated dose of AU-011 / laser applications from Cohorts 1 to 3 administered weekly for 2 treatments
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser
- Cohort 5 AU-011 & Laser (Experimental): AU-011/laser applications from Cohorts 1 to 3 administered weekly for 3 treatments. Up to 2 cycles of this regimen may be administered and subjects have the option of receiving a third cycle of treatment.
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser
- Cohort 6 AU-011 & Laser (Experimental): High dose of AU-011/laser applications administered weekly for 3 treatments and up to 3 cycles of treatment.
  Interventions: Drug: AU-011; Device: Suprachoroidal Microinjector; Device: PDT Laser

INTERVENTIONS:
Drug: AU-011 — AU-011 Via Suprachoroidal Administration
Device: Suprachoroidal Microinjector — Suprachoroidal Injection Device
Device: PDT Laser — Laser Administration

SUMMARY:
The primary objective is to determine the safety, tolerability, and preliminary efficacy of belzupacap sarotalocan for the treatment of primary indeterminate lesions and small choroidal melanoma (IL/CM).

DETAILED DESCRIPTION:
This is an open-label, ascending single and repeat dose escalation trial designed to evaluate the safety, tolerability, and preliminary efficacy of up to 4 dose levels and repeat dose regimens of belzupacap sarotalocan via suprachoroidal administration with 1 or 2 laser applications per treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary indeterminate lesion or small choroidal melanoma (IL/CM)
* Have no evidence of metastatic disease confirmed by imaging
* Be treatment naïve for IL/CM

Exclusion Criteria:

* Have known contraindications or sensitivities to the study drug or laser
* Active ocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Treatment related AEs and treatment related serious adverse events (SAEs). | 52 weeks
  Adverse Events

SECONDARY OUTCOMES:
Within-subject difference of historical tumor thickness growth rate and post-treatment growth rate over 52 weeks. | 52 weeks
  Tumor Thickness Growth Rate
Time to reach tumor progression | 52 weeks
  Tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences
Locations (22):
- United States (22):
  - Retina Associates SW, P.C., Tucson, Arizona
  - UCLA Jules Stein Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - UCHealth Eye Center, Aurora, Colorado
  - Retina Associates of Florida, Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - University of Illinois At Chicago Illinois Eye and Ear Infirmary, Chicago, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - University of Iowa Department of Ophthalmology and Visual Sciences, Iowa City, Iowa
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W. K. Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Associated Retinal Consultants, PC, Royal Oak, Michigan
  - Retina Center, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University Casey Eye Institute, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - St. Thomas Health / Tennessee Retina, PC, Nashville, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - University of Wisconsin Dept of Ophthalmology & Visual Sciences, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aura Biosciences — http://www.aurabiosciences.com/